CLINICAL TRIAL: NCT06812962
Title: A Pilot RCT on the Feasibility of an Online Quiz Game to Promote Tobacco-related Knowledge, Attitudes and Behaviours Among Primary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Principle investigator and associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: coshdrama2324
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Students will engage in an online quiz competition for 4 weeks on tobacco-related topics. Each day, students could answer a maximum of 5 questions.
  Interventions: Other: Online quiz competition
- Control (Active Comparator): Students will engage in an online quiz competition for 4 weeks on healthy eating-related topics. Each day, students could answer a maximum of 5 questions.
  Interventions: Other: Online quiz competition

INTERVENTIONS:
Other: Online quiz competition — The intervention and control students participated in an online quiz game on tobacco and healthy eating topics, respectively. Each day, students could answer a maximum of 5 questions randomly selected from the respective pool of questions by the platform. The students logged onto the online platform and played the quiz competition on weekdays for 4 weeks (i.e. total of 20 days).

SUMMARY:
The goal of this pilot RCT is to test the feasibility of an online quiz game to promote tobacco-related knowledge, attitudes and behaviours in local primary 5-6 school students. The main question it aims to answer is:

* Feasibility of intervention
* Acceptance of intervention by schools, teachers, parents and teachers
* Adherence to the 4-week intervention
* Functional online quiz platform
* Satisfaction of students and parents towards intervention Researchers will compare the questionnaire results from students to see if students doing tobacco-related questions on the online quiz platform will have better tobacco-related knowledge, higher anti-tobacco attitudes and lower intention to smoke.

Students will engage in an online quiz competition for 4 weeks on tobacco-related topics for the intervention group and on healthy eating for the control group. They will complete pre-test and post-test questionnaires before and after the online quiz competition.

ELIGIBILITY:
Inclusion Criteria:

* Primary 5-6 students from local primary schools
* Able to read and communicate in Chinese
* Have a digital device for online access to the quiz game at home

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 921 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | During the post-questionnaire at 5th-6th weeks and during the phone interview at 10th-16th weeks.
  Students and parents will be asked their comments towards intervention in the phone interview: [Students] 1) Did you find the quiz platform interesting or engaging? Why? 2) On a scale of 0 to 10, how much did you enjoy using the quiz platform? [Parents] 1) Do you think using a quiz competition format increases your child's motivation to learn? 2) Are there specific features or functionalities you think would enhance the platform for both parents and students? Students will be asked 'Do you think the interface of the online quiz competition platform is easy to use?' We will measure the number of times that the website developer or the students reported technical problems.
  We will also measure the participation rate of students during the online quiz competition period.

SECONDARY OUTCOMES:
Effectiveness of intervention on tobacco-related knowledge (including ASPs) | During the pre-questionnaire right before the intervention and post-questionnaire at 5th-6th weeks.
  Students reported their opinions towards 5 statements in pre and post tests: [Pre-test] 1) Tar causes addiction; 2) Exposure to secondhand smoke increases the risk of cancer; 3) The harm from e-cigarettes is less than that of traditional cigarettes; 4) Tobacco companies use various flavours to attract children to use e-cigarettes; 5) The Hong Kong government has already banned the sale of heated tobacco products. [Post-test] 1) Occasional smoking is harmless to health; 2) Exposure to secondhand smoke increases the risk of death; 3) E-cigarettes contain carcinogens; 4) Tobacco companies promote heated tobacco products through social media platforms; 5) The Hong Kong government has already banned the sale of e-cigarettes. All the statements have 5 options from definitely no to definitely yes. The options were recoded, as appropriate, with higher scores indicating knowing more about the harms and misleading marketing strategies of ASPs.
Effectiveness of intervention on tobacco-related attitudes (including ASPs) | During the pre-questionnaire right before the intervention and post-questionnaire at 5th-6th weeks.
  Students will report their opinions towards 5 statements: 1) Smokers are more stylish; 2) Adults should have the freedom to smoke in their homes; 3) Using e-cigarettes can bring a bit of enjoyment; 4) Tobacco companies have a contribution to society; 5) The government should implement a total ban on smoking. All the statements have 5 options from definitely no to definitely yes. The options will be recoded, as appropriate, with higher scores indicating knowing more about the harms and misleading marketing strategies of ASPs.
Effectiveness of intervention on tobacco-related intentions (including ASPs) | During the pre-questionnaire right before the intervention and post-questionnaire at 5th-6th weeks.
  Students were asked: If one of your good friends offers you an e-cigarette or heated tobacco product, ask you to have a few puffs, and no one will know about this as no more smoking in the future. Will you use them? There will be 5 options from definitely no to definitely yes.
Effectiveness of intervention on SHS and THS exposure at home | During the pre-questionnaire right before the intervention and post-questionnaire at 5th-6th weeks.
  Students were asked: In the past 7 days, how many days (0-7) 1) was someone smoking next to you when you were at home? 2) do you smell secondhand smoke drifting in from outside when you were at home? 3) was someone smoking next to you when you were outside home? 4) you can smell cigarette smoke on objects or people when you are at home and no one is smoking, and you don't see any smoke?
Effectiveness of intervention on tobacco use | During the pre-questionnaire right before the intervention and post-questionnaire at 5th-6th weeks.
  Students were asked: 1) Which of the following tobacco products have you ever used? 2) In the past 30 days, which of the following tobacco products have you used?

CONTACTS AND LOCATIONS:
Locations (1):
- Local primary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No